CLINICAL TRIAL: NCT03022734
Title: A Phase II Study of Neoadjuvant Systemic Chemotherapy With Short Course Radiotherapy in Patients With Unresectable Rectal Cancer and Liver Metastasis
Brief Title: Short Course Radiotherapy, Unresectable Rectal Cancer, Liver Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sang Joon Shin, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0410
Record Dates: First submitted 2017-01-10; First posted 2017-01-16 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Rectal Cancer, Metastatic
MeSH Terms: conditions — Rectal Neoplasms; Neoplasm Metastasis | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemotherapy with radiotherapy (Experimental): Cetuximab or Bevacizumab, FOLFOX or FOLFIRI, radiotherapy
  Interventions: Drug: chemotherapy; Radiation: radiotherapy

INTERVENTIONS:
Drug: chemotherapy — cetuximab 250mg/m2 or bevacizumab 5mg/kg, FOLFOX (oxaliplatin 85mg/m2, leucovorin 200mg/m2, 5-FU 400mg/m2, 5-FU continuous 1200mg/m2) or FOLFIRI (irinotecan 180mg/m2, leucovorin 200mg/m2, 5-FU 400mg/m2, 5-FU continuous 1200mg/m2)
Radiation: radiotherapy — After FOLFOX 4cycle, subject have short course radiotherapy 5Gy for 5 days.

SUMMARY:
The purpose of this study is the increase of resection rate of primary cancer in rectal after short course radiotherapy without interrupt chemotherapy schedule during the period of chemotherapy. Radiation therapy is followed by additional chemotherapy to prevent the progression of systemic metastasis, and to reduce the incidence of rectal carcinoma including metastasis.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed for unresectable (impossible to try Total mesorectal excision) rectal cancer with liver metastasis
* over 19 years
* Eastern Cooperative Oncology Group 0-1
* Proper organ function
* more than one target lesion (standard by Response Evaluation Criteria in Solid Tumors 1.1)
* Who should sign on the Informed consent form before participate the trial.

Exclusion Criteria:

* Metastasis in other organ except liver
* Chronic active hepatitis or cirrhosis
* History of treatment for metastatic colorectal cancer
* Subject pregnant or breast feeding
* Uncontrolled disease
* Have had adjuvant therapy
* Uncontrolled peripheral nerve infection
* Alcoholic or drug addict
* Subject currently is enrolled in or ≤30 days from ending other clinical trial.
* History of other type of cancer except resolved from skin cancer and cervical cancer.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
complete resection (R0) rate for rectal and liver lesions | after surgical resection, an average of 24 weeks

SECONDARY OUTCOMES:
Response rate (RECIST V1.1) | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No